CLINICAL TRIAL: NCT07124390
Title: Electroacupuncture as a Treatment for Refractory Overactive Bladder: A Pilot Randomized Controlled Trial
Brief Title: Electroacupuncture as a Treatment for Refractory Overactive Bladder
Acronym: EAOAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Principal Investigator, Elmas, Pelvic Health Physiotherapist, Chelsea and Westminster NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OAB; IRAS No: 1011199 (Other: HRA)
Record Dates: First submitted 2025-07-31; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Over Active Bladder; Urinary Incontinence (UI); Nocturia
Keywords: Electric-Acupuncture; Acupuncture; PTNS; Neuromodulation
MeSH Terms: conditions — Urinary Incontinence; Nocturia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: 3 arm parallel RCT
Who Masked: Participant, Investigator
Masking Description: PI will be blinded to randomisation and data collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Electroacupuncture (EA) Group Experimental (Experimental): Arm 1: Electroacupuncture (EA) Group Arm Type: Experimental Description: Participants in this group will receive electroacupuncture treatment targeting sacral and lower abdominal acupuncture points traditionally used for overactive bladder (OAB). Sterile, single-use acupuncture needles will be inserted and connected to an electroacupuncture device that delivers a low-frequency electrical current.
  Duration: 12 weekly sessions over 12 weeks Setting: Delivered by trained pelvic health physiotherapists in an outpatient hospital setting.
  Intervention:
  Interventions: Device: Name: Electroacupuncture (EA) Type: Device-based acupuncture therapy
- Arm 2: Percutaneous Tibial Nerve Stimulation (PTNS) Group (Active Comparator): Arm Type: Active Comparator Description: Participants in this group will receive percutaneous tibial nerve stimulation, a standard treatment for OAB. A fine needle electrode is inserted near the ankle to stimulate the tibial nerve, transmitting signals to the sacral nerve plexus that controls bladder function.
  Duration: 12 weekly sessions over 12 weeks Setting: Delivered by trained clinicians in an outpatient setting.
  Interventions: Device: Neuromodulation therapy
- Arm 3: Sham Acupuncture (Control) Group (Sham Comparator): Description: Participants in this group will receive non-penetrating sham acupuncture using blunt-tipped placebo needles that mimic the look and feel of real acupuncture but do not penetrate the skin or provide electrical stimulation. This is used as a control to assess the true efficacy of EA compared to placebo.
  Duration: 12 weekly sessions over 12 weeks Setting: Delivered by trained physiotherapists using standardised placebo protocols.
  Interventions: Device: Sham Acupuncture

INTERVENTIONS:
Device: Name: Electroacupuncture (EA) Type: Device-based acupuncture therapy — Description: Insertion of acupuncture needles at specific points with electrical stimulation (2 Hz) for 30 minutes per session.
  Arms: Arm 1: Electroacupuncture (EA) Group Experimental
Device: Neuromodulation therapy — Type: Neuromodulation therapy
  Description: Insertion of a needle electrode near the medial malleolus with low-voltage electrical stimulation (20 Hz) applied for 30 minutes per session.
  Other Names: Percutaneous Tibial Nerve Stimulation (PTNS)
  Arms: Arm 2: Percutaneous Tibial Nerve Stimulation (PTNS) Group
Device: Sham Acupuncture — Type: Placebo
  Description: Non-invasive, non-penetrating placebo needles placed at the same points as in the EA group, without electrical stimulation, for 30 minutes per session.
  Arms: Arm 3: Sham Acupuncture (Control) Group

SUMMARY:
Brief Summary

The goal of this clinical trial is to learn whether electroacupuncture (EA) is as effective and acceptable as percutaneous tibial nerve stimulation (PTNS) in treating overactive bladder (OAB) in adult women. The main questions it aims to answer are:

Does electroacupuncture reduce OAB symptoms to a similar extent as PTNS? Is electroacupuncture an acceptable and accessible treatment option for women with OAB?

Researchers will compare EA and PTNS with a third group receiving sham acupuncture to see whether EA offers similar or better symptom relief and is more acceptable to participants.

Participants will:

Be randomly assigned to one of three groups: EA, PTNS, or sham acupuncture

Receive one treatment session per week for 12 weeks

Complete symptom diaries, quality-of-life questionnaires, and feedback on treatment acceptability

Attend follow-up assessments after treatment ends

The study will take place at Chelsea and Westminster NHS Foundation Trust, with support from the hospital's Physiotherapy and Urology departments. It is funded by the Chelsea and Westminster Hospital Joint Research Committee (JRC) and Supported by Imperial Collage London.

DETAILED DESCRIPTION:
Detailed Description of the Study Background and Rationale Overactive bladder (OAB) is a chronic condition affecting millions of individuals worldwide, characterised by urinary urgency, frequency, nocturia, and in many cases, urge urinary incontinence. The condition has a significant impact on quality of life, including physical discomfort, emotional distress, social isolation, and increased risk of falls and infections in older adults. The prevalence of OAB is estimated to affect approximately 12-19% of adults in the UK, with similar prevalence globally. Despite this high prevalence, treatment options remain limited, with pharmacological agents often associated with side effects such as dry mouth, constipation, and cognitive impairment, particularly in older adults. Consequently, non-pharmacological treatments, including neuromodulation techniques, have gained attention.

Percutaneous tibial nerve stimulation (PTNS) is a well-established, minimally invasive neuromodulation technique that has demonstrated efficacy for OAB symptoms and is currently offered in some NHS settings. However, PTNS requires weekly clinic visits for a minimum of 12 weeks, making it resource-intensive and inaccessible for many patients, particularly those in underserved or rural communities.

Electroacupuncture (EA) is a promising alternative. EA involves the application of a mild electrical current to acupuncture needles inserted at specific anatomical points. Emerging evidence suggests that EA may modulate bladder function through neuromodulatory mechanisms similar to PTNS. EA has been used in traditional Chinese medicine for urological and gynaecological conditions and is increasingly recognised in Western medicine. Preliminary studies and systematic reviews have demonstrated potential benefits of EA for OAB symptoms, but the evidence is limited by small sample sizes, methodological weaknesses, and lack of control groups.

This randomised controlled trial (RCT) aims to provide high-quality evidence comparing the effectiveness and cost-effectiveness of electroacupuncture versus PTNS and sham acupuncture in the treatment of OAB in adult women.

Study Design

This is a three-arm, single-blind, randomised controlled trial. A total of 60 adult female participants with a clinical diagnosis of OAB will be recruited and randomised into one of three groups:

* Group 1: Electroacupuncture (EA)
* Group 2: Percutaneous Tibial Nerve Stimulation (PTNS)
* Group 3: Sham acupuncture (placebo control) Each group will consist of 20 participants. Randomisation will be computer-generated and stratified by age and baseline symptom severity.

The intervention period will last for 12 weeks. Participants will receive weekly 30-minute sessions of their allocated treatment during this period. Outcomes will be assessed at baseline, at the end of the 12-week intervention, and at 3-month follow-up.

Aim of the Proposed Study

Specific Aims

1. Assess whether the study can be delivered as planned.
2. Estimate the average (mean) scores and variability (standard deviation) of the primary outcome at baseline, after 12 weeks of treatment, and at 6- and 12-month follow-up.
3. Evaluate whether all elements of the study process - such as recruitment, randomisation, and data collection - work together smoothly.
4. Feasibility and Acceptability: I aim to test the feasibility of delivering EA in physiotherapist-led group settings and evaluate its acceptability and adherence among patients.
5. Clinical Outcomes: I will assess whether EA can reduce symptoms such as urinary urgency, frequency, and pelvic pain using validated measures.
6. Cost-Effectiveness: I will explore EA's suitability as a scalable and affordable alternative to PTNS and medications.

   Assessment and management of risk While both electroacupuncture and PTNS are low-risk interventions, potential side effects may include localised discomfort or minor bleeding. All participants undergoing treatment will be monitored by their treating physiotherapist as part of routine clinical care. Including those in the control group receiving sham EA, will be provided with a named contact and telephone number for support in the event of any concerns.

   All adverse events (AEs) and serious adverse events (SAEs) will be reported to the Research Ethics Committee and the SSG. A SAE is defined as any untoward medical occurrence that results in hospitalisation, is life-threatening, or results in significant distress directly related to the intervention.

   Primary Objective

   Aim:

   To determine whether electroacupuncture (EA) is as effective or more effective than percutaneous tibial nerve stimulation (PTNS) for reducing overactive bladder (OAB) symptoms, measured by validated patient-reported outcomes.

   Hypotheses:
   * Null Hypothesis (H0): EA has no difference in effectiveness compared to PTNS in reducing OAB symptoms.
   * Alternative Hypothesis (H1): EA is superior to PTNS in reducing OAB symptoms.

   PICOT Framework:
   * P - Adults diagnosed with OAB and/or urgency urinary incontinence (UUI).
   * I - Electroacupuncture (EA) delivered at the tibial nerve site.
   * C - Standard PTNS treatment (active control) and sham EA (placebo control).
   * O - Reduction in OAB symptoms (urgency, frequency, nocturia, incontinence) measured by ICIQ-OAB and bladder diary.
   * T - Outcomes assessed at baseline, mid-treatment (6 weeks), post-treatment (12 weeks), and follow-up at 6 and 12 months.

   Secondary Objectives
   * Assess the feasibility and acceptability of delivering EA in a physiotherapy-led clinical setting.
   * Evaluate recruitment, randomisation, treatment adherence, and data collection processes.
   * Estimate mean scores and variability (SD) of primary and secondary outcomes at each assessment point.
   * Explore the cost-effectiveness of EA compared to PTNS.
   * Assess impact on quality of life (QOL) domains including sleep, anxiety, and emotional well-being.

   Outcome Measures/Endpoints All selected measures are validated, patient-centred, sensitive to change, and minimise participant burden. Completion of all outcome measures at each assessment point is expected to take no more than 60 minutes at baseline and less at follow-ups.

   Demographic Data will be collected:

   Age, gender, ethnicity, religion, duration/nature of symptoms, previous treatments, occupation, education, socioeconomic status (postcode proxy).

   Primary Endpoint/Outcome Measurement Variable Participant-Level Metric Method of Aggregation Timepoints ICIQ-OAB total score (urgency, frequency, nocturia, incontinence) Change from baseline Mean change per group Baseline, 6 weeks, 12 weeks, 6 months, 12 months 3-Day Bladder Diary (episodes per 24h) Change from baseline Mean change per group Baseline, 6 weeks, 12 weeks, 6 months, 12 months Patient-Specific Functional Scale (PSFS) Change from baseline Mean score per group Baseline, 6 weeks, 12 weeks, 6 months, 12 months

   Secondary Endpoints/Outcomes Measurement Variable Participant-Level Metric Method of Aggregation Timepoints ICIQ-OABqol total and subdomain scores Change from baseline Mean score per group Baseline, 6 weeks, 12 weeks, 6 months, 12 months Visual Analogue Scale (VAS) for Pain Change from baseline Mean score per group Baseline, 6 weeks, 12 weeks, 6 months, 12 months Feasibility metrics (recruitment rate, retention, adherence) Proportions Rates and proportions Throughout study

   Exploratory Endpoints/Outcomes
   * Association between baseline patient characteristics (e.g., duration of symptoms, socioeconomic status) and treatment response.
   * Exploratory analysis of sleep and anxiety improvements using subdomains of ICIQ-OABqol.

   Table of Endpoints/Outcomes The following table summarises the primary, secondary, and exploratory outcome measures for this study. Outcome measures have been carefully selected through consultation with patients and specialist pelvic health physiotherapists to ensure they are clinically meaningful, validated, sensitive to change, and minimise participant burden. Each measure is mapped against the study objectives and corresponding assessment timepoints to provide a clear overview of data collection and evaluation throughout the trial.

   Objectives Outcome Measures Timepoint(s) of Evaluation Primary Objective ICIQ-OAB total score (symptom severity) 3-Day Bladder Diary Patient-Specific Functional Scale (PSFS) Baseline, 6 weeks, 12 weeks, 6 months, 12 months Secondary Objectives ICIQ-OABqol (quality of life) VAS for pelvic pain Feasibility metrics (recruitment, adherence, retention) Baseline, 6 weeks, 12 weeks, 6 months, 12 months Exploratory Objectives Association of baseline characteristics with outcomes Sleep and anxiety improvements (from ICIQ-OABqol subdomains) Baseline, 6 weeks, 12 weeks, 6 months, 12 months

   TRIAL SETTING This trial will be conducted at a single site: the Pelvic Health Physiotherapy Outpatient Department at Chelsea and Westminster Hospital NHS Foundation Trust.

   Participants will be recruited from patients referred to the outpatient pelvic health physiotherapy service who have completed a standard course of pelvic floor physiotherapy (3-6 months) for overactive bladder without satisfactory improvement.

   Typically, these patients are discharged back to their referring general practitioner or urogynaecology team for secondary care assessment.

   Before discharge, eligible patients will be invited to participate in the trial.

   Site-specific details:
   * All trial procedures (screening, consent, treatment delivery, and follow-up) will occur at Chelsea and Westminster Hospital.
   * No additional recruitment sites or Participant Identification Centres (PICs) are planned.
   * Recruitment will prioritise inclusion of patients from diverse socioeconomic and ethnic backgrounds to promote equity, access, and generalisability of findings.

   Practitioner eligibility:

   Only qualified pelvic health physiotherapists and acupuncture-trained practitioners with appropriate certifications and clinical experience will deliver the interventions.

   The usual care pathway in the NHS (physiotherapy first, then secondary care review if physiotherapy fails) will be maintained to reflect real-world practice and ensure pragmatic trial conditions.

   TRIAL PROCEDURES Aim Intervention Group 1: PTNS, Intervention Group 2: EA Control Group: Sham EA will mimic real EA and PTNS procedures but will use non-penetrating or minimal stimulation techniques at a site near, but not directly on, the tibial nerve.

   Participants in all groups will experience similar procedures, ensuring blinding is maintained.

   By incorporating a sham EA arm, this study ensures that any observed differences in treatment outcomes are due to the true physiological effects of electroacupuncture, rather than psychological or non-specific treatment effects.

   Key Notes:
   * Screening: After final physiotherapy appointment if symptoms persist. Screening and eligibility check occur before baseline.
   * Baseline Visit (Visit 1): Collection of baseline data, randomisation, and start of intervention scheduling.
   * Treatment Visits: Participants attend weekly outpatient sessions (up to 12 sessions total) depending on protocol assignment. Adverse event reporting will be monitored each visits.
   * Midpoint Check (Week 6): ICIQ-OAB questionnaire repeated to monitor progress.
   * Follow-up Visit (Months 6 and 12): Final outcome measures, , and collection of patient diaries.
   * Missed Treatments: If a session is missed, it can be rescheduled within the following 7 days if possible.

   Recruitment Participants will be identified at their final pelvic health physiotherapy appointment if their symptoms have not improved after at least three months of physiotherapy.

   Eligible patients will be invited to participate and provided with a Participant Information Sheet. An Introducer (a trained member of the team) will discuss the study, answer any questions, confirm eligibility, and seek written consent to schedule an outpatient appointment.

   Participants will not be eligible if they have a definite contraindication to treatment, judged against the eligibility criteria via a standardised screening procedure.

   Participants' GPs will be informed about their participation (with the patient's consent).

   Data about participants who are screened but not randomised (for CONSORT reporting) will include:
   * Age
   * Gender
   * Ethnicity (if applicable)
   * Registration/randomisation status Who will confirm eligibility? Eligibility will be confirmed by clinical staff directly involved in the participant's care (physiotherapists and urogynecologists).

   Note: If this were a CTIMP (Clinical Trial of an Investigational Medicinal Product), confirmation would need to be by a medical doctor, but in this non-CTIMP study, clinical confirmation is sufficient.

   Sample Size and Statistical Analysis A sample of 60 participants (20 per group) provides sufficient power to detect clinically meaningful differences in OABSS, assuming a non-inferiority margin of 3 points, a standard deviation of 3.5, 80% power, and a 5% significance level.

   Analysis will follow the intention-to-treat principle. ANCOVA will be used for primary outcome analysis adjusting for baseline scores. Pairwise comparisons between groups (EA vs PTNS, EA vs sham) will be conducted. Missing data will be handled using multiple imputation methods. A health economic analysis using QALYs will also be performed.

   Consent The Principal Investigator (PI) holds overall responsibility for research conduct at site, including obtaining informed consent. The PI will ensure that any individual delegated to obtain consent is authorised, trained, and competent, following the approved protocol, Good Clinical Practice (GCP) standards, and the Declaration of Helsinki (World Medical Association, 2013).

   Informed consent will be obtained before participants undergo any trial-specific procedures outside standard care, including the collection of identifiable data. Participants will be informed that they have the right to refuse participation without explanation. They may withdraw from the trial at any time without affecting their future care. Data and samples collected before withdrawal will be used only if prior consent for this has been given; this will be explained in the participant information materials.

   Should re-consent or new information arise, the PI is responsible for timely communication with participants. Vulnerable participants must be protected from coercion or undue influence.

   Where participants cannot read, write, or speak English, alternative consent processes will be used, including:
   * Use of witnesses for consent signing
   * Translated information sheets
   * Hospital interpreters (face-to-face or telephone services)
   * Verified AI translations checked by native speakers Consent documents will comply with GCP, local regulations and will be approved by the Research Ethics Committee (REC) before use.

   Participants will have opportunities to ask questions in person, by phone, or via email.

   Simple randomisation with a 1:1 allocation ratio will be used in this pilot study. Each participant will have an equal chance of being assigned to either treatment group. Simple randomisation prevents allocation bias and ensures unpredictability (Schulz and Grimes, 2002).

   Blinding Participants will be blinded to the treatment group - they will not know whether they are receiving PTNS, EA, or sham EA. However, due to the nature of the treatments, it will not be possible to blind the physiotherapists delivering the interventions. This limitation is common in trials of complex interventions (Roland & Torgerson, 1998; Stephenson & Imrie, 1998).

   Emergency Unblinding In this pilot study, participants may be unblinded if a valid medical or safety reason arises, such as pregnancy, diagnosis of active cancer, pacemaker insertion, or any other new contraindication to the intervention.

   Participants will be asked at each visit about any new diagnoses or symptoms to ensure they remain eligible to continue.
   * Code break responsibility: The randomisation codes will be securely held by the Principal Investigator (PI).

   Baseline Data Baseline data will be collected at the participant's initial visit prior to randomisation to ensure eligibility, allow group comparisons, and provide essential information for analysis.

   Trial assessments

   Assessments will take place in an outpatient physiotherapy clinic. Baseline assessment of participants will be made following written consent to participate in the Study.

   Assessments will be recorded on a standard sheet, manually and electronically and will comprise patient-reported outcome measures. Assessment sheets will be stored locally in locked cabinets and password-protected computers. Implementing a robust data management plan, conducting regular audits, and use secure storage will minimise the risk for data bridging.

   Outcome Measures Completion of all outcome measures is expected to take a maximum of 60 minutes at baseline (including demographic data), and a shorter time at follow-up(s).

   Demographic Data:

   Demographic data (age, gender, duration of symptoms, nature of symptoms, previous treatments, occupation, ethnicity, religion, gender, and socioeconomic status, like occupation, education, and post code will be collected to describe participant characteristics.

   The selection of both primary and secondary outcome measures for this study has been informed through patient and clinician engagement during the study's development phase. Consultations with patients living with overactive bladder (OAB) and urgency urinary incontinence (UUI), as well as with specialist pelvic health physiotherapists, helped to identify outcome measures that are clinically meaningful and relevant to patient experience and well-being. The overarching aim was to minimise participant burden while ensuring comprehensive and validated data collection across the most relevant domains of OAB impact (Donovan et al., 1996; Milsom et al., 2009). All tools selected are validated, widely used in pelvic health research, and have demonstrated sensitivity to change in similar populations.

   All necessary permissions have been obtained to use the International Consultation on Incontinence Questionnaire modules in this research.

   Long-term Follow-up Assessments Participants will be monitored after the active treatment phase through scheduled follow-up appointments.
   * Frequency of Follow-up Visits:

   Follow-up will occur at 6 months and 12 months after randomisation. These will be conducted either by telephone consultation or face-to-face (F2F) depending on the participant's preference.

   • Duration of Follow-up Appointments: Each follow-up consultation is expected to take approximately 45 minutes.

   • Assessments to be Carried Out:

   All Outcome Measures (OCMs) used at baseline will be repeated at each follow-up, including:
   * Symptom questionnaires
   * Medical history updates
   * Assessment of any new contraindications
   * Adverse event reporting • Difference from Standard Care: The follow-up visits and assessments are specific to the research study and are additional to standard care. In routine clinical practice, such structured and detailed follow-up would not be conducted at these intervals.

     • Retention Strategies:
   * Flexible options for follow-up (phone or F2F)
   * Reminder calls, texts, or emails ahead of scheduled visits
   * Clear communication about the importance of follow-up
   * Offering appointment flexibility around participant schedules • Definition of Lost to Follow-up: Participants will be considered 'lost to follow-up' if they miss two consecutive follow-up attempts (phone or F2F) and do not respond to further contact efforts (e.g., telephone, email, letter).

     * Measures for Missed Visits or Data Points:

   If a participant misses a scheduled follow-up, the research team will attempt:
   * Phone or email contact within 1 week of the missed appointment
   * Offering a re-arranged visit or telephone call
   * If necessary, collecting key outcomes via a brief telephone questionnaire • Outcome Data from Protocol Non-Adherers:

   Data will continue to be collected from participants even if they:
   * Deviate from the assigned treatment
   * Discontinue active treatment This ensures that outcome analysis includes all participants according to the intention-to-treat principle.

   Statistical Analysis Plan

   Baseline comparability will be assessed across randomised groups using the following variables:
   * Demographic data: age (continuous, mean ± SD), gender (categorical, %), ethnicity (categorical, %)
   * Clinical characteristics: duration of OAB symptoms (continuous), presence of comorbidities (categorical), baseline bladder diary metrics (continuous), and pelvic floor muscle function (ordinal via Oxford scale)
   * Psychosocial data: baseline anxiety and quality of life scores (continuous) Descriptive statistics will be presented as means and standard deviations or medians and interquartile ranges (IQRs), depending on data distribution. Categorical variables will be reported as frequencies and percentages. A CONSORT flow diagram will summarise participant progression through each stage of the trial.

   Primary Outcome Analysis The primary outcome is change in OAB symptom severity from baseline to 12 weeks, assessed via the Overactive Bladder Questionnaire Short Form (OAB-q SF).
   * Summary measures: Mean difference (with 95% confidence intervals) between groups at 12 weeks
   * Method of analysis: An independent t-test (if data is normally distributed) or Mann-Whitney U test (if non-normally distributed) will be used to compare change scores between the two arms.
   * Repeated measures approach: A mixed-effects linear model will also be used to account for within-subject variability across time points (baseline, week 6, week 12).
   * Handling of missing data: Multiple imputation methods will be employed to address missing primary outcome data, assuming data are missing at random. Sensitivity analyses will test the robustness of assumptions.
   * Subgroup analyses: Exploratory subgroup analyses will examine outcomes by age group, menopausal status, and baseline symptom severity.
   * Analysis population: All analyses will follow the intention-to-treat (ITT) principle. Per-protocol analyses will be conducted as secondary.
   * Qualitative data: A subset of participants will take part in qualitative interviews to explore treatment acceptability. These will be analysed thematically using NVivo.

   Secondary Outcome Analysis

   Secondary outcomes include:
   * Patient global impression of improvement (PGI-I)
   * Health-related quality of life (EQ-5D-5L)
   * Adverse events
   * Health service use (for economic analysis)

   Where appropriate:
   * Continuous outcomes will be analysed using independent t-tests or mixed-effects models.
   * Categorical outcomes (e.g. PGI-I categories) will be compared using chi-square or Fisher's exact tests.
   * Confidence intervals will be presented in preference to p-values, and secondary analyses will be interpreted as hypothesis-generating.

   Subgroup Analyses

   Pre-specified subgroup analyses will be conducted to explore differences in treatment effect by:
   * Age (<50 vs ≥50 years)
   * Baseline symptom severity (mild/moderate vs severe)
   * Prior exposure to conservative OAB therapies Interaction terms will be included in mixed models to assess treatment effect modification.

   Adjusted Analysis

   Adjusted analyses will be conducted for the primary and secondary outcomes to control for baseline imbalances and potential confounders, including:
   * Age
   * Baseline OAB symptom severity
   * Pelvic floor function score Continuous variables will be modelled as linear covariates. Adjusted and unadjusted results will both be reported, with the adjusted model considered the main analysis.

   Interim Analysis and Criteria for Premature Termination No formal interim efficacy analysis is planned due to the pilot nature of the study. However, a safety review will be conducted after the first 20 participants complete treatment to assess adverse events.

   This review will be conducted by an independent clinician and statistician not involved in the trial. If unexpected serious adverse events attributable to treatment occur in ≥10% of participants in either arm, the Chief Investigator will consult with the Sponsor and the Trial Steering Committee (TSC) to consider early termination. The trial team will remain blinded unless unblinding is deemed essential for safety decisions.

   Participant Population

   Three analysis populations will be defined:
   * All-randomised (ITT): All participants randomised, regardless of treatment receipt.
   * All-treated: Participants who received at least one session of the allocated intervention.
   * Per-protocol: Participants who received at least 9 of 12 planned treatment sessions and completed all outcome assessments.

   The primary analysis will use the ITT population. Safety analyses will use the all-treated population.

   Procedures to Account for Missing or Spurious Data

   To minimise missing data:
   * Participants will receive reminders via phone/email for outcome assessments.
   * Follow-up calls will be used to complete missed questionnaires.

   For analysis:
   * Reasons for missing data will be recorded.
   * Multiple imputation will be applied for the primary outcome and main secondary measures.
   * Sensitivity analyses will include:

     * Complete case analysis
     * Best-worst and worst-best case imputation for primary outcome

   Other Statistical Considerations Any deviations from this pre-specified statistical analysis plan will be documented and justified in the final study report. A separate statistical analysis plan (SAP) will be developed prior to database lock.

   If funding allows, a cost-effectiveness analysis (CEA) will be conducted using trial data to estimate incremental cost per QALY gained from the NHS perspective.

   Economic Evaluation A cost-utility analysis will be performed comparing EA and PTNS using EQ-5D-5L-derived utilities. Health resource use will be recorded using a patient-completed health service utilisation log. Costs will be derived from standard NHS tariffs. Results will be reported as incremental cost-effectiveness ratios (ICERs) and presented using cost-effectiveness acceptability curves (CEACs).

   DATA MANAGEMENT

   Data will be collected via paper case report forms (CRFs) and then entered into a secure, validated electronic database. Source documents include hospital records, clinic letters, bladder diaries, and signed informed consent forms. CRFs will include:

   All source documents and signed consent forms will be stored in secure, locked cabinets at the trial site and archived per regulatory requirements.

   Data Handling and Record Keeping

   Data will be handled according to GCP and NHS Trust data governance policies:

   All data will be anonymised before analysis. At the end of the trial, data will be archived securely for 10 years in accordance with Trust and regulatory requirements.

   Access to Data Direct access to trial data will be granted to authorised representatives of the Sponsor, Chelsea and Westminster NHS Foundation Trust, the host institution, and the relevant regulatory authorities to facilitate trial-related monitoring, audits, and inspections. This access will be in accordance with participant consent and applicable data protection legislation. Only personnel authorised by the Chief Investigator will be permitted access to the final trial dataset.

   Research Ethics Committee (REC) Review & Reports The trial will be conducted in compliance with the UK Policy Framework for Health and Social Care Research and will be approved by a Research Ethics Committee (REC) prior to initiation.

   The protocol, informed consent documents, participant-facing materials (e.g., advertisements, GP letters), and any substantial amendments will be submitted for REC approval. Substantial amendments will not be implemented until a favourable opinion is received from the REC, and, where applicable, approvals from the MHRA and NHS R&D departments are also obtained.

   All REC-related correspondence will be retained in the Trial Master File (TMF) and Investigator Site Files (ISFs).

   The Chief Investigator will be responsible for:
   * Submitting Annual Progress Reports (APR) within 30 days of the REC approval anniversary
   * Notifying the REC of the End of Trial, including reasons for early termination if applicable
   * Submitting a Final Report within 12 months of trial completion, including study results and any relevant publications or conference abstracts

   Peer Review This trial has undergone proportionate, independent, expert peer review in accordance with NIHR Clinical Research Network (CRN) standards to ensure scientific and methodological quality.
   * Independence: The trial protocol was reviewed by at least two experts independent of the investigators' host institution and not involved in any aspect of the study.
   * Expertise: Reviewers had subject-matter expertise in pelvic health, physiotherapy-led interventions, clinical trials, and acupuncture-related methodologies.
   * Proportionality: As a single-centre, three-arm feasibility study (EA vs PTNS vs sham acupuncture), the level of peer review was appropriate to the trial's size and complexity.

   Details of the peer review process are documented and available upon request from the Sponsor or Chief Investigator.

   Public and Patient Involvement (PPI) Patients and members of the public have been actively involved in the design and planning of this trial. A pelvic health Patient and Public Involvement (PPI) representative contributed to the development of the research question, intervention acceptability, and the design of patient-facing materials.

   The trial aligns with INVOLVE guidance on PPI and demonstrates a commitment to meaningful involvement throughout the research lifecycle.

   Dissemination Results from this trial will be disseminated in line with Good Clinical Practice (GCP) and relevant ethical standards. Data will be owned by Chelsea and Westminster Hospital NHS Foundation Trust and the Chief Investigator (CI). A final trial report will be prepared following CONSORT guidelines and made available via clinical trial registries and on request.

   Investigators may publish secondary analyses with prior written approval from the CI and sponsor. All publications will be reviewed to ensure consistency, with a minimum 30-day review period. No unnecessary embargoes will be applied.

   All outputs will acknowledge funding sources and contributors. Participants will be offered a lay summary of the results, and individual results may be requested via the Principal Investigator after study completion.

   The trial protocol, final report, anonymised dataset, and statistical code will be shared publicly post-publication, under controlled access agreements and in compliance with data protection regulations.

   Funding and Support Partial funding for the study is provided by the Chelsea and Westminster Hospital's Continuing Professional and Clinical Development (CPCD) programme. Applications are pending for additional funding from charitable research trusts and internal NHS innovation funds.

   The study is led by a pelvic health physiotherapist with academic supervision from a university research mentor and oversight by a multidisciplinary advisory group including experts in acupuncture, urogynaecology, trial methodology, and statistics.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

* Female adults aged 18 years or older.
* Diagnosed with overactive bladder syndrome (ICIQ-OAB score ≥10).
* Symptoms present for at least three months and refractory to first-line treatments.
* Willing to refrain from starting new bladder-related treatments during the study period.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Participants meeting any of the following criteria will be excluded:

  * Pregnant or planning pregnancy during the study period.
  * Bleeding disorders.
  * Severe needle phobia.
  * Presence of a pacemaker.
  * Active cancer diagnosis.
  * Active urinary tract infections or other urological conditions requiring urgent intervention.
  * Participation in another clinical trial for bladder dysfunction within the past six months.
  * Neurological conditions affecting continence (e.g., diabetic neuropathy, multiple sclerosis, Parkinson's disease).
  * Life-threatening infections.
  * Severe cognitive deficits, unconsciousness, dementia (e.g., Alzheimer's or other neurodegenerative diseases).
  * History of incontinence surgery.
  * Previous acupuncture for OAB within the past two months.
  * History of thromboses.
  * Recovering from or suffering from a serious illness or major surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified genders eligible to participate:
  Women (Cisgender women)
Enrollment: 60 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Improvement in Overactive Bladder Symptoms Using the International Consultation on Incontinence Questionnaire - Overactive Bladder Module (ICIQ-OAB) | This questionnaire will be completed at 6 weeks, 12 weeks, 6 months, and 12 months
  Participants will complete the validated International Consultation on Incontinence Questionnaire - Overactive Bladder (ICIQ-OAB) at baseline, 6 weeks, 12 weeks, 6 months, and 12 months to assess changes in urinary symptoms, including urgency, frequency, nocturia (waking up to urinate), and incontinence.
  The ICIQ-OAB is a standardised, reliable, and responsive patient-reported outcome measure commonly used to monitor the severity and impact of overactive bladder symptoms. It consists of four symptom-specific questions, each scored from 0 to 4 or 0 to 5, resulting in a total score range from 0 to 16, where higher scores indicate more severe symptoms.
  A decrease in total score over time will indicate an improvement in OAB symptoms. The measure is sensitive to change, making it appropriate for tracking the effectiveness of interventions over multiple time points.
Change in Urinary Frequency and Incontinence Episodes via 3-Day Bladder Diary | This questionnaire will be completed at 6 weeks, 12 weeks, 6 months, and 12 months
  Participants will complete a bladder diary for 3 consecutive days at baseline, 6 weeks, 12 weeks, 6 months, and 12 months. This diary captures frequency of voids, incontinence episodes, urgency, and fluid intake. Bladder diaries are a gold standard for tracking urinary behaviour and treatment response in OAB management. Less visit to toilet will show positive outcome
Change in Functional Activity Measured by Patient-Specific Functional Scale (PSFS) | This questionnaire will be completed at 6 weeks, 12 weeks, 6 months, and 12 months
  Participants will identify up to three daily activities affected by overactive bladder (OAB) and rate their ability to perform each activity on a scale from 0 to 10, using the Patient-Specific Functional Scale (PSFS). A score of 0 indicates they are unable to perform the activity at all, while a score of 10 reflects their prior or normal level of function before symptoms began.
  The PSFS is a patient-centred, valid, and responsive measure that allows individuals to report the specific functional limitations that matter most to them. This personalised approach ensures relevance and sensitivity to change, as it captures the real-life impact of OAB on daily functioning.
  An increase in scores over time will indicate an improvement in function and reduced symptom interference, while stable or declining scores may suggest limited benefit or worsening symptoms. This tool complements symptom-based questionnaires by focusing on individual goals and quality of life.

SECONDARY OUTCOMES:
The International Consultation on Incontinence Questionnaire - Overactive Bladder Quality of Life (ICIQ-OABqol) will be used to assess the impact of overactive bladder (OAB) symptoms on participants' quality of life. | This questionnaire will be completed at 6 weeks, 12 weeks, 6 months, and 12 months
  This validated questionnaire evaluates key domains such as emotional wellbeing, social embarrassment, sleep disruption, and coping strategies, providing a comprehensive view of how OAB affects daily living.
  Each domain is scored on a scale where higher scores indicate greater negative impact and poorer quality of life. By tracking scores over time, the study will assess whether interventions lead to improvements in quality of life. A reduction in scores from baseline will indicate a positive response to treatment, suggesting reduced symptom burden and better psychosocial outcomes.
  This tool is sensitive to change and widely used in both clinical and research settings to evaluate the real-world effects of OAB and its management.
Pain Intensity Measured by Visual Analogue Scale (VAS) | This questionnaire will be completed at 6 weeks, 12 weeks, 6 months, and 12 months
  Participants will rate their pain intensity in the bladder and legs. The VAS is a validated and widely used tool for assessing pain, where participants mark a point on a 10 cm line ranging from 0 (no pain) to 10 (worst imaginable pain).This outcome measure will help monitor any discomfort potentially associated with the treatments, electroacupuncture (EA) or percutaneous tibial nerve stimulation (PTNS). By comparing scores across time points and treatment groups, researchers can identify whether either intervention leads to increased, decreased, or unchanged levels of musculoskeletal pain.
  Lower VAS scores over time would indicate reduced pain and improved comfort, while higher scores may suggest adverse effects or worsening symptoms. Including multiple pain intensities (current, least, worst) provides a more nuanced understanding of the participants' pain experience.
Patient Satisfaction Assessed by Likert-Scale Questionnaire | This questionnaire will be completed at 12 weeks
  Participants will complete a Likert-scale-based questionnaire co-designed with patient input to measure satisfaction, perceived benefit, and overall treatment experience. It will be administered after the final treatment session (12 weeks).
  he tool uses a series of 5-point Likert scale items (e.g., strongly disagree to strongly agree) to capture participants' views on various aspects of the treatment process, including:
  How satisfied they were with the treatment
  Whether they perceived any improvement in their symptoms
  How easy or burdensome the treatment was to follow
  Whether they would recommend the treatment to others Higher scores will indicate more positive experiences and greater satisfaction, helping to inform future service delivery and identify areas for improvement
Incremental Cost-Effectiveness Ratio (ICER) of EA vs. PTNS | This questionnaire will be completed at 12 months
  Cost-effectiveness will be evaluated using ICER to compare the cost per unit improvement in symptom severity and quality-adjusted life years (QALYs) between EA and PTNS. Economic data will be collected throughout treatment and follow-up.
Frequency and Severity of Adverse Events | From beginning of trial to 12 months after the trial
  All adverse events related to EA or PTNS will be recorded and categorised by severity and causality. Monitoring will follow ICH Good Clinical Practice (E6[R2]) standards to ensure participant safety.
Treatment Compliance and Attendance Rates | From randomisation to 12 weeks after randomisation
  Participant adherence will be tracked through a treatment log. Missed sessions and reasons for non-attendance will be recorded to assess treatment feasibility and refine delivery strategies for future implementation.
Long-Term Symptom and Functional Outcomes at 6 and 12 Months | will be completed at, 6 months, and 12 months
  Participants will be followed up at 6 and 12 months via telephone or face-to-face appointments. All outcome measures taken at the beginning of trial will be repeated. This extended assessment will evaluate sustainability of treatment effects and any delayed responses.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Professor Regan, Study Chair — Obstetrics and Gynaecology and Consultant in Gynaecology at the Imperial College and Consultant at NHS Trust St Mary's Hospital Campus; Deepa Dr Abichandani, Study Chair — Senior Lecturer in Physiotherapy Employability Lead for School of Allied and Community Health London South Bank Universit; Mark Pro. Johnson, Study Chair — Senior Lecturer, Consultant in Obstetrics and Obstetric Medicine Charing Cross Hospital. And Chelsea and Westminster NHS Trust Imperial College London Clinical Chair in Obstetrics Department of Metabolism, Digestion an; Rufus Mr. Cartwright, Study Director — Uro-gynaecologist consultant and Honorary Clinical Senior Lecturer institute of Reproductive and Developmental Biology, Hammersmith Campus and Celsea and Westminster NHS Trust Gynaecology and Departm; Elmas X Court, Principal Investigator — Chelsea and Westminster Hospital and Imperial College London
Locations (1):
- Chelsea and Westminster hospital NHS foundation Trust, London, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available

REFERENCES:
- See also: not available at present — https://www.researchgate.net/publication/392078318_Needling_the_Urge_A_New_Solution_for_Pelvic_Control_RCT_trial